CLINICAL TRIAL: NCT01514552
Title: A Pilot Phase I Study of the Use of Functional Confections in Promoting Oral Health in Men and Women
Brief Title: The Use of Functional Confections in Promoting Oral Health
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Yael Vodovotz, Associate Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2010H0073
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Oral Health; Oral Cancer; Gum Disease
Keywords: Functional food; Strawberries; Gummies; Smoker; Nonsmoker
MeSH Terms: conditions — Mouth Neoplasms; Gingival Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo gummy (Placebo Comparator): Each 6 gram placebo gummy contains 79% corn syrup (Karo, ACH Food Companies, Memphis, TN), 20% wheat starch (Confectioners G, Tate and Lyle PLC., Decatur, IL), 1% artificial strawberry flavors (Kool-Aid Kraft Foods, East Hanover, NJ).
  Interventions: Other: Placebo control gummy
- Strawberry gummy (Active Comparator): Each 6 gram strawberry gummy contains 45% freeze-dried fruit (California Strawberry Commission), 44% corn syrup (Karo, ACH Food Companies, Memphis, TN), 11% wheat starch (Confectioners G, Tate and Lyle PLC., Decatur, IL). With this formulation, daily fruit consumption is equivalent to 1 cup of whole strawberries. All ingredients (wheat starch, freeze-dried fruit, and high fructose corn syrup) will be purchased from a single lot. When a single lot is not available then the multiple manufacturing lots will be mixed into a single lot to be used for production of fruit gummies.
  Interventions: Other: Strawberry gummy

INTERVENTIONS:
Other: Strawberry gummy — Randomized to consume 2 gummies (6 gram gummies each, total 12 grams/dose)four times daily for 7 days. Subjects will be randomized to either start with this strawberry intervention during intervention days 0 to 7 or during the crossover intervention on days 21 to 28.
  Arms: Strawberry gummy
Other: Placebo control gummy — Randomized to consume 2 gummies (6 gram gummies each, total 12 grams/dose)four times daily for 7 days. Subjects will be randomized to either start with this a placebo gummy intervention during intervention days 0 to 7 or during the crossover intervention on days 21 to 28.
  Arms: Placebo gummy

SUMMARY:
In areas of the world where populations are undernourished poor oral health is prevalent. Diets rich in fruit and vegetables are thought to have many health benefits including reducing the risk of oral cancer or gum disease. In particular fruits such as strawberries contain many different compounds which may be responsible for these proposed health benefits.

From this study, the researchers hope to gain information about how the tissues in the mouth absorb strawberry gummies in a population of habitually smoking and never smoking men and women. The researchers will measure inflammation hormones in your saliva and urine and the genes in your mouth and blood. Two different strawberry gummies will be tested in this study. The strawberry gummies were developed at OSU in the Department of Food Science and Technology. One type of strawberry gummy will contain freeze-dried whole strawberries while the other type will have no fruit. In total the eight pieces of strawberry gummies that you will consume in one day will be at most equal to 1 cup of whole strawberries. The research team believes the two strawberry gummies may be digested and absorbed differently and that components in the strawberry gummies may be helpful for oral health.

DETAILED DESCRIPTION:
Polyphenols (plant chemicals, some produce purple and red color in fruits) found in strawberries have been associated with reducing the risk of gum disease. However, much of these chemicals are susceptible to degradation during food processing and digestion. Minimally degraded in the mouth, polyphenols when consumed as fresh fruits are retained only for brief periods. Therefore, exposure of fresh fruit polyphenols to oral tissues may not be adequate for a biologic effect to occur. At OSU, food scientists have developed a 6 gram strawberry gummy containing 3 grams of freeze-dried strawberries designed to dissolve relatively slow in the mouth.

The investigators will investigate the effects of strawberry gummy consumption on oral health in 36 habitually smoking and non-smoking healthy adults (men and women). At the enrollment visit (Day-14), subjects will visit the OSU Clinical Research Center (CRC) for an oral brushing; submit a 24-hour urine collection, and a saliva sample. Subjects will then start an anthocyanin-free (avoid purple and red fruits and vegetables) diet which they will maintain for 6 weeks of this study. After 2 weeks, subjects will have their first "washout" visit at the CRC. This visit will be one of two "washout visits" where subjects will again submit samples (fasting blood, urine, saliva, and oral brushing). At this visit, smokers will be block randomized (random assignment using computer software) into one of two groups (strawberry or placebo gummies) with a matching non-smoker having the same gender and age group. A salivary pharmacokinetic (sPK) study will follow and involves collection of saliva at these time points: 5 minutes before gummy placed in the mouth, and at 5,10,15,20,25, and 30 minutes after gummies have been in the mouth. Subjects will be instructed to consume 2 pieces of strawberry, or placebo gummy 4 times a day for 7 days. After 7 days subjects return to the CRC for a "treatment visit" to submit fasting blood, urine, saliva and oral brushing samples. Subjects will repeat the two-week anthocyanin-free diet and return to the CRC for another "washout visit" before crossing over to the other study gummy. After 7 days of gummy consumption, subjects will return for their second treatment visit and submit fasting blood, oral brushing, saliva, and 24 hour urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Submit to a 24 hour urine cotinine test which will be used to determine smoking status.
* Meet one of the following smoking criteria

Non-smoker

* Does not currently smoke or has no history of smoking or using tobacco related products (cigarettes, cigars, pipe, snuff, or chewing tobacco) or smoking any non-tobacco related products and urine cotinine (less than 100 ng/mL
* Does not currently smoke but has quit smoking for more than 10 years and smoked less than 1 pack/day of cigarettes when they were actively smoking and has a urine cotinine (less than 100 ng/mL).

Smoker

* Smokes habitually at least 10 cigarettes/day and a urine cotinine level of >1000 ng/mL. Cigar and pipe smokers who smoke at least 10 grams of tobacco daily are also eligible.
* Agree to consume a standardized vitamin and mineral supplement and avoid other nutritional, dietary, or alternative medications/supplements for the duration of the study.
* No history of malabsorptive, gastrointestinal or other metabolic disorders requiring special diet recommendations.
* Body mass index (BMI) between 20 and 35 kg/m2
* Abstain from purple and red colored foods and beverages which contain significant anthocyanins and polyphenols
* Abstain from the use of ANY mouth washes (commercial or home remedies)during 6 week study period

Exclusion Criteria

* Have a known allergy to strawberries, corn, and wheat products or those who have never consumed any of these products.
* Have active metabolic or digestive illnesses such as malabsorptive disorders (Crohn's, ileus, IBS), renal insufficiency, hepatic insufficiency, hyper- or hypothyroidism, cachexia, morbid obesity, or short bowel syndrome.
* Have a history of pituitary hormone diseases that currently require supplemental hormonal administration (thyroid hormones, ACTH, growth hormone, insulin) or other endocrine disorders requiring hormone administration.
* Have significant loss of gastrointestinal organs due to surgery, except for appendix.
* Have altered immunity such as chronic inflammatory disease, autoimmune disorders, cancer, anemia, hemophilia, and blood dyscrasias.
* Heavy alcohol consumers defined as >15 glasses/week (one glass = 1.5 oz. liquor, 5 oz. wine, or 12 oz. beer).
* Antibiotic use in the last 6 months or on medications that will accelerate or decrease bowel motility.
* Are receiving or in need of dental treatment during the study period.
* Have noticeable open lesions, sores that have not healed for more than 3 months, have had any active oral lesions or maladies within the last month, or have a history of leukoplakia, tumors of the buccal cavity, throat, and lips.
* Have difficulty swallowing (dysphagia), pain with swallowing (odynophagia), salivary gland dysfunction, or xerostomia (dry mouth).
* A "non-smoker" who is currently or has a history (less than 10 years of smoking abstinence) of either tobacco or non-tobacco related smoking.
* Women, who are planning to conceive in the next 6 months, suspect they are pregnant, pregnant, or nursing.
* Are taking medications that inhibit clotting (warfarin sodium) or using prescribed oral rinses (Peridex).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-11; Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Achieve excellent compliance and minimal toxicity with consumption of the strawberry gummies. | one week after intervention
  Daily records of consumption will be maintained. Standardized qualitative and quantitative toxicity criteria (NIH Common Terminology Criteria for Adverse Events, v. 3.0) will be employed to describe the safety as well as incidence toxicity

SECONDARY OUTCOMES:
Quantify the enteral absorption and excretion patterns of strawberry polyphenols in smoking and non-smoking healthy adult men and women consuming the strawberry and placebo gummies. | Day 0, 7, 21, and 28
  This data will be used to define relationships between dietary intake, polyphenol metabolism and the biological outcomes examined in tertiary outcome.
  1. Pharmacokinetics of strawberry polyphenols in saliva following consumption of a single dose delivering two 6 gram fruit gummies will be compared in smoking and non-smoking men and women consuming the strawberry or placebo gummies.
  2. Prevalent strawberry polyphenols and their metabolites in saliva, serum, and urine will be assessed and compared with strawberry gummy type consumed.
Measure salivary inflammatory markers and gene expression profiles in oral mucosa that promote oral health following short-term exposure to strawberry fruit polyphenol. | Day 0, 7, 21, 28
  1. Salivary inflammatory markers (cortisol, Ig A, and 8-hydroxydeoxyguanosine) following consumption of strawberry and placebo gummies will be compared in smoking and non-smoking men and women.
  2. Expression profiling will be examined on RNA obtained from longitudinal buccal brushings and plasma utilizing qRT-PCR and SuperArray's RT2 Profiler™ PCR Array (Inflammation Panel) containing 84 genes unique to the inflammation pathway and compared with strawberry gummy type consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Vodovotz, PhD., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States